CLINICAL TRIAL: NCT03237273
Title: HEAD-US SCORING SYSTEM: Assessment of the Real-world Impact of Ultrasound on Disease Management and Treatment Decision-making in Moderate and Severe Haemophilia
Brief Title: HEAD-US SCORING SYSTEM: Assessment of the Real-world Impact of Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 63143
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Moderate and Severe Haemophilia
MeSH Terms: conditions — Lymphoma, Follicular; Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): All patients will undergo ultrasound scan using the HEAD-US Scoring System by a non-imaging specialist
  Interventions: Other: HEAD-US scoring system

INTERVENTIONS:
Other: HEAD-US scoring system — HEAD-US scoring system - Ultrasound scan performed by a non-imaging specialist to assess for joint bleed or damage

SUMMARY:
Ultrasound represents a promising technique for the assessment of joint health in persons with haemophilia (PWH) by non-imaging specialists. The Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) programme has been developed with the aim of integrating joint ultrasound in the routine assessment of PWH through the use of a simplified scoring system. The inter-operator reliability of the technique among European haemophilia treaters has been validated and described elsewhere. Further work is needed to assess the real-world impact of ultrasound on disease management and treatment decision-making.

DETAILED DESCRIPTION:
Patients are seen routinely in clinic by specialist haemophilia physiotherapists who assess the patients using the Haemophilia Joint Health Score tool (HJHS). Trial participants will be seen during their routine clinic visits and will be seen by a clinician and the physiotherapist who will carry out the routine assessment along with the HEAD-US scan.

Patients will be seen a maximum of 4 times throughout the year from registration of the first patient, according to their visit schedule, but will only be scanned at the first visit.

Results will be analysed to determine if the treatment decision-making is influenced by the results of the scan

ELIGIBILITY:
Inclusion Criteria:

* Moderate (FVIII/FIX:C 1-5%) and severe (FVIII/FIX: C <1%) patients with haemophilia A or B aged ≥ 6 years
* On demand or prophylaxis treatment regimen

Exclusion Criteria:

* Joints with a previous history of surgery
* Joints with damage as a result of causes other than haemophilia-related bleeding

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Any change in treatment | 12 months
  Any change in treatment including, management of a bleed and/or change in routine treatment protocol (including changes to prophylaxis regimen, or decision to start/stop prophylaxis regimen) as a result of the ultrasound findings

SECONDARY OUTCOMES:
% joints with normal HJHS and abnormal HEAD-US score | 12 months
  % joints with normal HJHS and abnormal HEAD-US score (for knees, ankles amd elbows separately
% joints with abnormal HJHS and normal HEAD-US score | 12 months
  % joints with abnormal HJHS and normal HEAD-US score

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Dolan, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
Data will be analysed and reported as results not individual data